CLINICAL TRIAL: NCT02658279
Title: A Proof-of-Concept, Pilot Study of Pembrolizumab (MK-3475) in Patients With Recurrent Malignant Glioma With a Hypermutator Phenotype
Brief Title: Pembrolizumab (MK-3475) in Patients With Recurrent Malignant Glioma With a Hypermutator Phenotype
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other); University of California, San Francisco (Other); Huntsman Cancer Institute/ University of Utah (Unknown); University of California, Los Angeles (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-227
Record Dates: First submitted 2016-01-12; First posted 2016-01-18 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Glioma; Recurrent Malignant Glioma
Keywords: Pembrolizumab (MK-3475); 15-227; Hypermutator Phenotype
MeSH Terms: conditions — Glioma | interventions — pembrolizumab

ARMS (1):
- Pembrolizumab (MK-3475) (Experimental): Pembrolizumab 200 mg will be administered as an approximately 30 minute (-5/+10 mins) IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. Patients will be followed with DCE perfusion MRI done at baseline and every 9 weeks (+/- 7 days). Patients will be allowed to stay on treatment in spite of increase in tumor size, provided the patient has no, or manageable, new neurologic symptoms, and at the discretion of treating physician. In that situation, tumor resection should be encouraged for the distinction between tumor progression and immunologic reactions. Patients undergoing surgical resection will have tissue collected for collateral studies. All collected tissue will be stored in the Pathology Core Tissue bank at MSK.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: (MK-3475)

SUMMARY:
The purpose of this study is to test if the study drug called pembrolizumab could control the growth or shrink the cancer but it could also cause side effects. Researchers hope to learn if the study drug will shrink the cancer by half, or prevent it from growing for at least 6 months. Pembrolizumab is an antibody that targets the immune system and activates it to stop cancer growth and/or kill cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant glioma by enrolling institution:

  * WHO grade IV tumors (GBM or its variants)
  * WHO grade III anaplastic astrocytoma or oligodendroglial tumors or
  * WHO grade II gliomas, if MRI shows contrast enhancement
* Tumor recurrence after previous treatment, which must have included at least radiation therapy and one cytotoxic chemotherapy. There is no limit on number of previous recurrences or lines of treatment.
* Previously obtained tumor sample exhibits a hypermutator phenotype. For the purposes of this trial, a hypermutator phenotype is defined as tumors harboring 30 mutations (non-synonymous somatic point or indel mutations) detected by the MSK-IMPACT or comparable next generation sequencing performed in a CLIA environment. Contingent to approval by the MSK Principal Investigator, patients with less than 30 mutations may be eligible if they display a mutation in a mismatch repair gene or other mutations in genes known to be associated with hypermutator phenotypes or microsatellite instability, including but not limited to MLH1, MSH2, MSH6, PMS2, POLE, POLD as determined by validated methods, or if microsatellite instability is present, as identified by polymerase chain reaction (PCR) or other validated methods.

  *Note: The MSK-IMPACT (Integrated Mutation Profiling for Actionable Cancer Targets) assay is a next generation genomic profiling performed on formalin-fixed, paraffin-embedded (FFPE) tumor tissue in a CLIA-certified Molecular Diagnostic Service laboratory. IMPACT provides full exon coverage of 410 cancer related genes and can detect base substitutions, small indels, copy number alterations and selected gene re-rearrangements. In some cases, additional assays such as Sanger Sequencing or fluorescence in situ hybridization (FISH) may be required to confirm specific results detected on IMPACT. Patients at MSK will have this assay to determine eligibility. Use of other validated next-generation sequencing techniques for eligibility may be considered, provided they are performed in a CLIA-certified laboratory and are approved by the MSK Principal Investigator.
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* An interval of ≥ 12 weeks from the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiation treatment field
* An interval of ≥ 4 weeks after the last administration of any investigational agent or any other treatment prior to first dose of pembrolizumab
* Must have recovered (i.e., ≤ Grade 1 or at baseline) from adverse events of any previous treatment. Note: Surgical resection for recurrent tumor prior to enrollment is allowed.
* Karnofsky performance status of ≥ 70
* Demonstrate adequate organ function as per below. All screening labs should be performed within 14 days of treatment initiation.

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Serum creatinine ≤1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
  * Albumin >2.5 mg/dL
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 9.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Subjects requiring escalating or chronic supraphysiologic doses of corticosteroids (> 10 mg/d of prednisone equivalent) for control of disease at the time of registration
* Previous or current treatment with an anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has a diagnosis of immunodeficiency, including Human Immunodeficiency Virus (HIV) or acquired immunodeficiency syndrome (AIDS)
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has a known history of active TB (Bacillus Tuberculosis)
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e.

with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Unable to undergo MRI of the brain (i.e. pacemaker or any other contraindication for MRIs).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has previously received treatment with bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
response rate | 1 year
  patients with stable disease will be considered responders if disease is stable for 27 weeks or more. The regimen will be considered worthy of further study if responses as defined above are observed in at least 3 of the 12 subjects. All subjects will undergo DCE-MRI of the head at the time points specified in Study Flow Chart . Local radiologic assessment of tumor measurements will be used during the study for clinical management and investigator-assessed disease progression. Additional MRIs may be obtained at the discretion of the investigators, as clinically indicated. Radiologic response (complete response or partial response) will be assessed by comparing on-treatment MRI scans with the pretreatment baseline MRI scans. Radiologic progression will be determined by using the smallest tumor measurement of either the pretreatment baseline or after initiation of study medication. The RANO criteria will be used for determining disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (16):
- United States (16):
  - University of California, Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Md Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/